CLINICAL TRIAL: NCT04135183
Title: Assessing Effectiveness of Community Acquired Pneumonia Treatment by Continuous Pneumonia Severity Score: a Prospective Observational Study and Randomized Controlled Trial
Brief Title: Assessing Effectiveness of Community Acquired Pneumonia Treatment by Continuous Pneumonia Severity Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I2019001440
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired Pneumonia; Pneumonia severity scores
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: This study consisting of two parts: the randomized controlled study include three groups, comprehensive evaluation group (traditional treatment group), PSI evaluation group and Expand-CURB evaluation group.The prospective observational study include one group. There are a total of 4 groups in the present study.
Masking Description: The present study is a randomized controlled open label trial. Patients and their physicians know the group and the treatment plan, and there are clear criteria for the final outcome (30-day fatality rate, length of stay). The masking is not required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comprehensive evaluation group (Experimental): The effectiveness of initial treatment and the next treatment plan were determined based on the CAP guidelines of Chinese Thoracic Society (CTS) or Infectious Diseases Society of America/American Thoracic Society(IDSA/ATS). The evaluation process was independently evaluated and documented by at least two clinicians. In case of disagreement, the final determination shall vote on the majority of votes.
  Interventions: Procedure: changes of Pneumonia Severity Score
- PSI evaluation group (Experimental): The changes of PSI scores and serum CRP were used to evaluate the therapeutic effects. If both PSI scores and CRP suggest that treatment is effective, the initial treatment will be maintained. If either of PSI scores or serum CRP suggest that treatment is effective, the initial treatment can be maintained, but need to be reviewed in the next 3-5 days. If both PSI scores and serum CRP suggest that the treatment is failed, the initial treatment should be changed. The change of initial treatment is not limited to antibiotics, but also include using glucocorticoid, ICU admission, mechanical ventilation according to the patients' condition.
  Interventions: Procedure: changes of Pneumonia Severity Score
- Expand-CURB evaluation group (Experimental): The changes of Expand-CURB scores and serum CRP were used to evaluate the therapeutic effects. If both Expand-CURB scores and CRP suggest that treatment is effective, the initial treatment will be maintained. If either of Expand-CURB scores or serum CRP suggest that treatment is effective, the initial treatment can be maintained, but need to be reviewed in the next 3-5 days. If both Expand-CURB scores and serum CRP suggest that the treatment is failed, the initial treatment should be changed. The change of initial treatment is not limited to antibiotics, but also include using glucocorticoid, ICU admission, mechanical ventilation according to the patients' condition.
  Interventions: Procedure: changes of Pneumonia Severity Score
- Prospective observational group (No Intervention): Patients' Expand-CURB scores, PSI scores and serum CRP before and after 3-5 days of initial treatment will be recorded. And the initial treatment, whether the initial treatment was changed 3-5 days of initial treatment and the final outcomes (ICU admission, 30-day mortality, average length of stay) will be recorded.

INTERVENTIONS:
Procedure: changes of Pneumonia Severity Score — assessing effectiveness of CAP treatment by using continuous pneumonia severity score
  Arms: Comprehensive evaluation group; Expand-CURB evaluation group; PSI evaluation group

SUMMARY:
Community acquired pneumonia (CAP) is a common respiratory infection and is the main cause of ICU admission and death in adults. Because of most patients were treated empirically against suspected causative microorganism, it is important to assess the effectiveness of treatment after 3 days of anti-infective therapy. However, the criteria for treatment failure is lack of a clear-cut and validated definition from the CAP guidelines.

Pneumonia severity scores is a wide-used severity rating system for treatment selection and outcome prediction for CAP. So far, the pneumonia severity scores only used once before the treatment started. Considering the pneumonia severity scores could reflect the severity of pneumonia, it is reasonable to assume that the change of pneumonia severity scores could reflect the patients' condition and the effectiveness of the treatment. This trail will be designed to validate the feasibility of assessing effectiveness of CAP treatment by using continuous pneumonia severity score.

DETAILED DESCRIPTION:
The applicant has established a CAP patients database and found a new effective pneumonia severity score: Expand-CURB. According to the retrospective study results, applicant found the changes of pneumonia severity score could reflect the patients'condition and was the independent risk factor for 30-day mortality. More specifically, if the patients'Expand-CURB score was not improved after 3-5 days of initial treatment, the odds ratio of 30-day mortality was 5.571 and 5.249 (95%CI 1.831-15.051, P=0.002) by univariate analysis and multivariate analysis (the multivariate was adjusted by the initial severity of pneumonia).

In addition, the applicant found the changes of serum CRP(C reactive protein ) before and after initial treatment also associated the patients'outcomes. If the serum CRP decreased less than 40% or not lower than 20mg/dl after the initial treatment, the odds ratio of 30-day mortality will be 3.692 and 3.806 (95%CI 1.867-7.756, P<0.001) by univariate analysis and multivariate analysis.

In conclusion, the applicant established three criteria for assessing effectiveness of CAP treatment:

1. Effective treatment by PSI: the PSI score decreased after 3-5 days the initial treatment.
2. Effective treatment by Expand-CURB: the Expand-CURB score decreased after 3-5 days the initial treatment.
3. Effective treatment by serum CRP: the serum CRP decreased more than 40% or lower than 20mg/dl after 3-5 days the initial treatment.

Furthermore, the applicant found combined pneumonia severity scores with CRP could predict the 30-day mortality more efficiently. The OR for both CRP and PSI treatment failure was 2.377 (95%CI 1.100-5.136, P=0.028). And the OR for both CRP and Expand-CURB treatment failure was 7.332 (95%CI 1.563-34.385, P=0.012). Therefore, it is reasonable to assume that the change of pneumonia severity scores and CRP could reflect the patients'condition and the effectiveness of the treatment.

To validate the feasibility of assessing effectiveness of CAP treatment by using continuous pneumonia severity score and changes of CRP, applicant intend to randomly allocate the patients into three arms: Comprehensive evaluation group, PSI evaluation group and Expand-CURB evaluation group. Patients who did not agree to participate the randomized controlled study will be asked whether they agree to provide their clinical data for prospective observational studies.

The primary outcomes will be 30-day mortality and ICU admission. The second outcome is length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* community acquired pneumonia(by CTS or IDSA/ATS guidelines)
* severe community acquired pneumonia(PSI scores >= 90 or Expand-CURB scores >= 4);

Exclusion Criteria:

* HIV patients
* Other immunodeficiency disorders (neutropenia, hematologic and solid tumors undergoing chemoradiotherapy, organ transplantation, and long-term treatment with glucocorticoid and cytokine antagonists).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients for ICU admission | through study completion, an average of 10 days
  Rate of patients who received ICU treatment during hospitalization. The numerator is the number of patients who received ICU treatment during hospitalization. The denominator is the number of all the enrolled patients.
Rate of all-caused mortality within 30 days. | through study completion, an average of 10 days
  Rate of all-caused death occurring within 30 days during hospitalization. The numerator is the number of patients who defined as death occurring within 30 days of hospitalization. The denominator is the number of enrolled patients.

SECONDARY OUTCOMES:
Length of stay for patients | through study completion, an average of 10 days
  The duration of a single episode of hospitalization. Inpatient days are calculated by subtracting day of admission from day of discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Fine MJ, Auble TE, Yealy DM, Hanusa BH, Weissfeld LA, Singer DE, Coley CM, Marrie TJ, Kapoor WN. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997 Jan 23;336(4):243-50. doi: 10.1056/NEJM199701233360402. PMID 8995086
- [Background] Liu JL, Xu F, Zhou H, Wu XJ, Shi LX, Lu RQ, Farcomeni A, Venditti M, Zhao YL, Luo SY, Dong XJ, Falcone M. Expanded CURB-65: a new score system predicts severity of community-acquired pneumonia with superior efficiency. Sci Rep. 2016 Mar 18;6:22911. doi: 10.1038/srep22911. PMID 26987602
- [Background] Welte T, Kohnlein T. Global and local epidemiology of community-acquired pneumonia: the experience of the CAPNETZ Network. Semin Respir Crit Care Med. 2009 Apr;30(2):127-35. doi: 10.1055/s-0029-1202941. Epub 2009 Mar 18. PMID 19296412